CLINICAL TRIAL: NCT02150746
Title: Circulating Tumor Cells Shed in Operative Blood During Pancreatectomy for Pancreatic Cancer is Responsible for Peritoneal Recurrence
Brief Title: Circulating Tumor Cells in Operative Blood
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-00271
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Pancreatic ductal adenocarcinoma; Pancreatic cancer; PDAC; Circulating tumor cells
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Buffy coat isolated from collected whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Cancer CTC: Peripheral/Central Venous Blood Draw Peritoneal Wash
  Interventions: Procedure: Peripheral/Central Venous Blood Draw; Procedure: Peritoneal Wash

INTERVENTIONS:
Procedure: Peripheral/Central Venous Blood Draw — Baseline sample of whole blood to be assessed for circulating tumor cells. Samples will be acquired via venipuncture unless a pre-existing central venous catheter is in place in which case the sample will be drawn from this.
Procedure: Peritoneal Wash — Prior to the start of the surgical resection, irrigation of the abdominal cavity will be performed and collected to determine baseline pancreatic cancer cells that may be present in the abdominal cavity.

SUMMARY:
It is hypothesized that circulating tumor cells (CTCs) from pancreatic adenocarcinoma are released into the peritoneal cavity through blood lost during the surgical resection of these tumors resulting in peritoneal recurrence despite appropriate surgical resection. Targeting the mechanisms responsible for CTC adhesion to the peritoneum may result in inhibition of implantation and growth, thus preventing this mode of pancreatic cancer recurrence postoperatively.

DETAILED DESCRIPTION:
Research Plan:

Intraoperative Subjects with Pancreatic Ductal Adenocarcinoma (PDAC) who have been consented and enrolled into the study will be taken to the operating room (OR) for their previously planned pancreatectomy procedure. After general anesthesia is induced, using universal precautions, blood sample (10ml) will be collected into a heparin tube for identification of circulating tumor cells (CTCs) and serve as one of two controls designed to assess background CTC counts. Once the participant has undergone surgical exploration as planned and has been deemed a candidate for resection, normal saline will be used to wash the abdominal cavity and collected in a suction canister by the attending surgeon. Abdominal washings are a normal part of the operative procedure, typically performed at the end of the operation to wash blood out of the abdominal cavity and is performed with variable amounts depending on the surgeon's discretion. For purposes of a control for the study, this wash step will be moved to the beginning of the operation. Additional washes/irrigations may be necessary at the end of the case at the surgeon's discretion. Cells collected in this fluid will be centrifuged and collected in the lab for determination of the presence of malignant cells. This will serve as the second of two controls. As the pancreatectomy procedure proceeds, subject blood will be lost as a normal consequence of the procedure and suctioned from the operative field into a new container containing heparin chilled on ice to preserve cell viability. This blood is normally discarded at the end of the case but a portion of the blood will be collected and utilized for downstream lab experiments to detect CTCs.

Laboratory/Post-Processing Blood collected in the operating room as described above will be immediately brought to the laboratory and centrifuged to separate out the plasma, buffy coat, and erythrocytes. The buffy coat, which contains the CTCs, white blood cells, and platelets, is removed and added to the commercially available cocktail per the kit protocol. Ficoll enrichment and separation of the CTCs will then be performed. The isolated CTCs will then be used for further downstream characterization and experimentation which will include, but not limited to: identification of CTC number, growth of CTCs in vitro and in vivo, and identification/characterization of CTC adhesion molecules which allow binding to human peritoneum. Any unused blood or component of blood not utilized in the experiment will be assigned a unique identifier and de-identified of patient for future cross-reference and stored at -80 degrees Fahrenheit at the University of Florida for potential future experiments or repeat CTC isolation.

Participant Data Collection On all enrolled subjects, the following de-identified information will be collected: participant demographic data, clinical and pathologic data, and data on cancer recurrence and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed tissue diagnosis of pancreatic ductal adenocarcinoma
* Scheduled to undergo pancreatectomy (open or minimally invasive) with curative intent
* Aged 18-85 years
* No race restrictions

Exclusion Criteria:

* Patients who have undergone preoperative therapy with either chemotherapy, radiation therapy, or both
* Serum CA19-9 less than 200ng/ml
* Patients with prior history of gastrointestinal malignancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-85 years with a confirmed tissue diagnosis of pancreatic ductal adenocarcinoma who are scheduled to undergo curative surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with isolated circulating tumor cells | 2 days
Percentage of patients with successful in vivo animal engraftment of isolated circulating tumor cells | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Thomas, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz MH, Wang H, Fleming JB, Sun CC, Hwang RF, Wolff RA, Varadhachary G, Abbruzzese JL, Crane CH, Krishnan S, Vauthey JN, Abdalla EK, Lee JE, Pisters PW, Evans DB. Long-term survival after multidisciplinary management of resected pancreatic adenocarcinoma. Ann Surg Oncol. 2009 Apr;16(4):836-47. doi: 10.1245/s10434-008-0295-2. Epub 2009 Feb 5. PMID 19194760
- [Background] Sugiura T, Uesaka K, Mihara K, Sasaki K, Kanemoto H, Mizuno T, Okamura Y. Margin status, recurrence pattern, and prognosis after resection of pancreatic cancer. Surgery. 2013 Nov;154(5):1078-86. doi: 10.1016/j.surg.2013.04.015. Epub 2013 Aug 22. PMID 23973112
- [Background] Katz MH, Pisters PW, Evans DB, Sun CC, Lee JE, Fleming JB, Vauthey JN, Abdalla EK, Crane CH, Wolff RA, Varadhachary GR, Hwang RF. Borderline resectable pancreatic cancer: the importance of this emerging stage of disease. J Am Coll Surg. 2008 May;206(5):833-46; discussion 846-8. doi: 10.1016/j.jamcollsurg.2007.12.020. Epub 2008 Mar 17. PMID 18471707
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Kuhara H, Eto K, Baba H. A proposal of a practical and optimal prophylactic strategy for peritoneal recurrence. J Oncol. 2012;2012:340380. doi: 10.1155/2012/340380. Epub 2012 Feb 8. PMID 22481921
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Yagi Y, Matsuda M, Yonemura Y, Baba H. Extensive intraoperative peritoneal lavage as a standard prophylactic strategy for peritoneal recurrence in patients with gastric carcinoma. Ann Surg. 2009 Aug;250(2):242-6. doi: 10.1097/SLA.0b013e3181b0c80e. PMID 19638909
- [Background] Cancer Facts & Figures 2013. Atlanta: American Cancer Society; 2013